CLINICAL TRIAL: NCT00030992
Title: A Phase II Clinical Trial of BMS-247550 (NSC 710428), an Epothilone B Analog, in Renal Cell Carcinoma
Brief Title: BMS 247550 to Treat Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Antonio T. Fojo, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020130; 02-C-0130; NCT00033670 (obsolete NCT alias)
Record Dates: First submitted 2002-02-20; First posted 2002-02-21 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-06

CONDITIONS: Renal Cell Carcinoma
Keywords: Epothilone B; Ixabepilone; Renal Cell Carcinoma; Kidney Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — ixabepilone; Ranitidine; Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-247550 (Experimental): One hour infusion on five successive days (daily x 5) every three weeks. Starting dose of 6 mg/m^2/day for a total per cycle dose of 30 mg/m^2
  Interventions: Drug: BMS-247550; Drug: Ranitidine; Drug: Diphenhydramine

INTERVENTIONS:
Drug: BMS-247550 — One hour infusion on five successive days (daily x 5) every three weeks. Starting dose of 6 mg/m^2/day for a total per cycle dose of 30 mg/m^2
Drug: Ranitidine — 50 mg 30-60 minutes prior to Ixabepilone (BMS-247550)
  Other Names: Zantac
Drug: Diphenhydramine — 50 mg intravenously 30-60 minutes prior to Ixabepilone (BMS-247550)
  Other Names: Benadryl; Diphenhist; Diphedryl

SUMMARY:
This study will examine whether the experimental drug BMS 247550 (Ixabepilone) is an effective treatment for kidney cancer. BMS 247550 belongs to a class of drugs called epothilones that interfere with the ability of cancer cells to divide. In the way they kill cells, they are very similar to a class of compounds known as the taxanes, which include the drug Taxol. Other characteristics of the epothilones, however, enable them to work in cells that are resistant to Taxol.

Patients 18 years of age or older with kidney cancer that has not spread to the central nervous system (unless the brain tumor has remained stable for at least six months after surgical or radiation treatment) may be eligible for this study. Pregnant or nursing women may not participate. Candidates are screened with various tests that may include blood and urine tests, electrocardiogram (EKG), and chest x-ray. Computerized tomography (CT) scans or X-rays, and possibly nuclear medicine studies may be done to determine the extent of disease.

Participants receive BMS 247550 by a 1-hour infusion into a vein for 5 consecutive days (days 1, 2, 3, 4 and 5) of each 21-day treatment cycle. Patients must stay in the National Institutes of Health (NIH) area near Bethesda, Maryland, for 7 to 8 days during the first treatment cycle and for the 5 days of treatment in subsequent cycles. The total number of cycles will vary among patients, depending on their individual clinical situation. The drug dose may be increased gradually in subsequent cycles in patients who can tolerate such increases. In addition, participants undergo the following tests and procedures:

* Periodic physical examinations and frequent blood tests
* X-ray and other imaging studies to determine if the tumor is responding to the treatment.
* Tumor biopsies to confirm the diagnosis or spread of tumor and to examine the reaction of certain proteins in cancer cells to BMS 247550. Two biopsies will be done. For this procedure, a small piece of tumor tissue is withdrawn through a needle under local anesthetic.

Treatment will be stopped in patients whose tumor grows while receiving BMS 247550. Patients whose tumor disappears completely will be followed at NIH periodically for examinations and tests. Patients whose disease does not completely resolve or whose disease recurs may be advised of other appropriate research protocols at NIH or, if none are available, will be returned to the care of their local doctor.

DETAILED DESCRIPTION:
Background:

BMS-247550 (NSC 710428), (ixabepilone) is a semi-synthetic analog of the natural product epothilone B.

The epothilones are a novel class of non-taxane microtubule-stabilizing agents obtained from the fermentation of the cellulose degrading myxobacteria, Sorangium cellulosum.

BMS-247550 is active against cancer models that are naturally insensitive to paclitaxel or have developed resistance to paclitaxel, both in-vitro and in-vivo.

Objectives

Establish the efficacy of the investigational agent BMS-247550 in patients with renal cell carcinoma when administered as a one hour infusion on day 1 to 5 every 21 days.

Evaluate the plasma pharmacokinetics of BMS-247550.

Explore the pharmacodynamics of BMS-247550 using an assay that measures the amount of endogenous tubulin in peripheral blood mononuclear cells (PBMC) that exists in the polymerized versus the unpolymerized state.

Determine the extent to which pharmacodynamic changes are observed over a range of doses of BMS-247550.

Determine if cross-resistance to BMS-247550 exists in patients who have previously received sorafenib or sunitinib.

Eligibility:

Age greater than 18.

Pathological confirmation of renal cell carcinoma.

Prior chemotherapy including sorafenib and sunitinib is allowed.

Design:

Phase II study.

BMS-247550 will be administered on days 1 through 5, every 21 days.

Restaging will be done every two cycles.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must fulfill all of the following criteria to be eligible for study admission:

1. Age greater than or equal to 18 years.
2. Histologic or cytologic confirmation of renal cell carcinoma (clear cell, type I and type II papillary, chromophobe, collecting duct and medullary).

   Patients should either:
   1. have received interleukin-2 (IL-2);
   2. have been evaluated for therapy with IL-2 and deemed to be ineligible; or (c) have been evaluated for therapy with IL-2 and refused treatment.
3. Measurable extent of disease.
4. Performance Status Eastern Cooperative Oncology Group (ECOG) 0-2.
5. Life expectancy of 3 months or greater.
6. Suitable candidate for receiving planned therapy as evidenced by screening laboratory assessments of hematologic, renal, hepatic, and metabolic functions:

   platelet count greater than or equal to 100,000/mL, absolute granulocyte count (AGC) greater than or equal to 1,500/mL, serum creatinine less than or equal to 1.6 or a measured creatinine clearance greater than or equal to 40 ml/min, serum glutamic pyruvic transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) less than or equal to 2.5 x normal limit (NL), and total bilirubin less than or equal to 1.5 x NL (in patients with clinical evidence of Gilberts' disease, less than or equal to 3 x NL).
7. Greater than or equal to 4 weeks from prior cytotoxic chemotherapy, radiation or immunotherapy; greater than or equal to 2 weeks from prior targeted-therapy (cytostatic agents); such patients should have recovered from toxicity from the prior therapy.
8. No serious intercurrent medical illness.
9. The ability to understand and willingness to sign a written informed consent form, and to comply with the protocol.
10. Patients should either: (a) have received sorafenib and or sunitinib and had progressive disease while receiving the drug(s) or (b) been intolerant to the drugs(s), or (c) been evaluated for therapy with sorafenib and or sunitinib and deemed to be ineligible; or (d) have been evaluated for therapy with sorafenib and or sunitinib and refused treatment.

EXCLUSION CRITERIA:

Patients with any of the following will be excluded from study entry:

1. Pregnant or nursing women are not eligible; neither are women or men of childbearing potential unless using effective contraception as determined by the patient's physician.
2. Patients with a history of central nervous system (CNS) metastases, because symptoms/signs of progressive disease may be confused with drug-related toxicities, unless control has been achieved with either radiation or surgical resection at least six months prior to enrollment on study.
3. Patients who are poor medical risk because of other non-malignant systemic disease or active, uncontrolled infection.
4. Human immunodeficiency virus (HIV) seropositive patients. Patients infected with the HIV virus will be excluded from this trial because the effect of BMS-247550 on HIV replication and/or the immune system is unknown and may be potentially harmful.
5. Prior craniospinal radiation, or total body irradiation (TBI).
6. Patients receiving other investigational drugs, or St. John's Wort (St. John's Wort can induce P450 and alter drug metabolism).
7. Common Toxicity Criteria (CTC) Grade 2 or greater motor or sensory neuropathy.
8. Known prior severe hypersensitivity reactions to agents containing Cremophor EL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2002-02; Primary Completion 2009-01 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tito Fojo, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wilson L, Jordan MA. Microtubule dynamics: taking aim at a moving target. Chem Biol. 1995 Sep;2(9):569-73. doi: 10.1016/1074-5521(95)90119-1. PMID 9383460
- [Background] Huizing MT, Misser VH, Pieters RC, ten Bokkel Huinink WW, Veenhof CH, Vermorken JB, Pinedo HM, Beijnen JH. Taxanes: a new class of antitumor agents. Cancer Invest. 1995;13(4):381-404. doi: 10.3109/07357909509031919. PMID 7627725
- [Background] Von Hoff DD. The taxoids: same roots, different drugs. Semin Oncol. 1997 Aug;24(4 Suppl 13):S13-3-S13-10. PMID 9335511
- [Result] Huang H, Menefee M, Edgerly M, Zhuang S, Kotz H, Poruchynsky M, Huff LM, Bates S, Fojo T. A phase II clinical trial of ixabepilone (Ixempra; BMS-247550; NSC 710428), an epothilone B analog, in patients with metastatic renal cell carcinoma. Clin Cancer Res. 2010 Mar 1;16(5):1634-41. doi: 10.1158/1078-0432.CCR-09-0379. Epub 2010 Feb 23. PMID 20179242
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2002-C-0130.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 102 participants were enrolled in this study.
Period: Overall Study
Arm/Group | BMS-247550
Started | 102
Completed | 102
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BMS-247550
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 79
  >=65 years | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 57.21 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 84
  African American | 12
  Asian | 5
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate is the percentage of participants with a response assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions, Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions,progressive disease (PD) is at least a 20% increase in the sum of the LD of target lesions or the appearance of one or more new lesions, stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 6 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | BMS-247550
Number analyzed (Participants) | 102
Percentage of participants
  Complete response | 1
  Partial Response | 9.4
  Progressive disease | 12.6
  Stable disease | 76.8

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 10 years
Measure: Number; unit: Participants
Arm/Group | BMS-247550
Number analyzed (Participants) | 102
Participants | 99

ADVERSE EVENTS:
Time Frame: 10 years
Arm/Group | BMS-247550
Serious Adverse Events (participants affected / at risk) | 40/102
Other Adverse Events (participants affected / at risk) | 99/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-247550 (N=102)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline phosphatase (Investigations) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Cardiac left ventricular function (Cardiac disorders) | 1 (1)
Cardiac troponin T (cTnT) (Cardiac disorders) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 1 (1)
Circulatory or cardiac-Other (hypertension) (Cardiac disorders) | 1 (1)
CNS cerebrovascular ischemia (Cardiac disorders) | 1 (1)
CPK (creatine phosphokinase) (Investigations) | 1 (1)
Creatinine (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 6 (6)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 5 (5)
Dysphagia, esophagitis, odynophagia (painful swallowing) (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Edema (General disorders) | 1 (1)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 3 (4)
Hemoglobin (hgb) (Blood and lymphatic system disorders) | 4 (4)
Hemoglobin increased (Investigations) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemorrhage/bleeding associated with surgery (Blood and lymphatic system disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 3 (3) — (documented clinically or microbiologically) with grade 3 or 4 neutropenia
Infection with neutropenia (Infections and infestations) | 1 (1)
Infection without neutropenia (Infections and infestations) | 7 (7)
Infection, Other (other than fever with neutropenia) (Infections and infestations) | 2 (2)
Joint, muscle, or bone (osseous)-Other (fracture) (Musculoskeletal and connective tissue disorders) | 1 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (3)
Neurologic-Other (autonomic neuropathy) (Nervous system disorders) | 2 (2)
Neuropathic pain (Nervous system disorders) | 1 (2) — e.g. jaw pain, neurologic pain, phantom limb pain, post-infectious neuralgia, or painful neuropathies
Neuropathy-motor (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 (5)
Pain-neuropathic (Nervous system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pericardial effusion/pericarditis (Cardiac disorders) | 1 (1)
Pulmonary-Other: malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure(s) (Nervous system disorders) | 1 (1)
SGOT (AST) (Investigations) | 1 (1)
SGPT (ALT) (Investigations) | 1 (1)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT (Infections and infestations) | 3 (3)
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Thrombosis/embolism (Vascular disorders) | 1 (3)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Voice changes/stridor/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2) — e.g. hoarseness, loss of voice, laryngitis
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 1 (1)
Fever (General disorders) | 8 (8) — in the absence of neutropenia, where neutropenia is defined as AGC< 1.0x109/L
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMS-247550 (N=102)
Fatigue (General disorders) | 13 (32)
Neuropathy-motor (Nervous system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 61 (76)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain or cramping (Gastrointestinal disorders) | 12 (19)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 4 (12)
Alanine aminotransferase increased (Investigations) | 3 (5)
Alkaline phosphokinase (Investigations) | 24 (33)
Alkaline phosphokinase increased (Investigations) | 4 (6)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 12 (16)
Allergic rhinitis (Immune system disorders) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 15 (19)
Allergy-Other (rhinitis) (Investigations) | 1 (1)
Amylase (Investigations) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 12 (52)
Anorexia (Metabolism and nutrition disorders) | 56 (88)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 31 (49)
Aspartate aminotransferase increased (Investigations) | 6 (13)
Bilirubin (Hepatobiliary disorders) | 6 (10)
Blood and lymphatic system disorders-Other, specify (bruising) (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Hepatobiliary disorders) | 4 (8)
Blurred vision (Eye disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Cardiac-ischemia/infarction (Cardiac disorders) | 1 (1)
Catheter-related infection (Infections and infestations) | 3 (3)
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 7 (9)
Chills (General disorders) | 2 (2)
Cholesterol high (Investigations) | 1 (1)
Circulatory or cardiac-Other (edema) (Cardiac disorders) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 30 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (39)
CPK (creatine phosphokinase) (Investigations) | 4 (5)
CPK increased (Investigations) | 2 (4)
Creatinine (Investigations) | 15 (21)
Creatinine increased (Investigations) | 5 (14)
Dehydration (Metabolism and nutrition disorders) | 16 (22)
Depressed level of consciousness (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis, focal (Skin and subcutaneous tissue disorders) | 1 (1) — associated with high-dose chemotherapy and bone marrow transplant
Diarrhea (Gastrointestinal disorders) | 4 (4)
Diarrhea (without colostomy) (Gastrointestinal disorders) | 42 (95)
Dizziness (Nervous system disorders) | 2 (2)
Dizziness/lightheadedness (Nervous system disorders) | 8 (9)
Dry eye (Eye disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2)
Dyspepsia/heartburn (Gastrointestinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dysuria (painful urination) (Renal and urinary disorders) | 1 (1)
Ear and labyrinth disorders-Other, specify (tinnitus) (Ear and labyrinth disorders) | 1 (1)
Edema (General disorders) | 14 (19)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) — (e.g. Stevens-Johnson syndrome, toxic epidermal necrolysis)
External auditory canal (Ear and labyrinth disorders) | 1 (1)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 3 (4)
Eye disorders-Other, specify (blepharitis) (Eye disorders) | 2 (2)
Fatigue (lethargy, malaise, asthenia) (General disorders) | 73 (220)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — fever of unknown origin without clinically or microbiologically documented infection
Fever (General disorders) | 2 (2)
Fever (in absence of neutropenia, where neutropenia is defined as AGC<1.0x109/L) (General disorders) | 30 (35)
Flushing (Vascular disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
GI-Other (bloating) (Gastrointestinal disorders) | 2 (2)
Headache (Nervous system disorders) | 15 (21)
Hematuria (Renal and urinary disorders) | 1 (1)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 6 (9)
Hemoglobin (hgb) (Blood and lymphatic system disorders) | 65 (235)
Hemoglobin increased (Investigations) | 1 (10)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hemorrhage/bleeding associated with surgery (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hot flashes/flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 12 (18)
Hypercholesterolemia (Investigations) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (28)
Hyperkalemia (Metabolism and nutrition disorders) | 15 (24)
Hypermagnesemia (Metabolism and nutrition disorders) | 6 (9)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 10 (13)
Hyperuricemia (Metabolism and nutrition disorders) | 9 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 62 (113)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (22)
Hypokalemia (Metabolism and nutrition disorders) | 9 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 19 (45)
Hyponatremia (Metabolism and nutrition disorders) | 18 (37)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (10)
Hypotension (Vascular disorders) | 6 (7)
Incontinence (Renal and urinary disorders) | 1 (1)
Infection without neutropenia (Infections and infestations) | 30 (41)
Infection, Other (skin) (Infections and infestations) | 8 (8)
Infections and infestations-Other, specify (skin) (Infections and infestations) | 4 (5)
INR increased (Investigations) | 4 (6)
Insomnia (Psychiatric disorders) | 13 (15)
Joint, muscle, or bone (osseous)-Other (myalgia) (Musculoskeletal and connective tissue disorders) | 4 (4)
Leukocytes (total WBC) (Investigations) | 34 (96)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 7 (30)
Lymphocyte count increased (Investigations) | 1 (1)
Memory loss (Nervous system disorders) | 1 (1)
Middle ear/hearing (Ear and labyrinth disorders) | 2 (2)
Mood alteration-anxiety agitation (Psychiatric disorders) | 3 (3)
Mood alteration-depression (Psychiatric disorders) | 8 (10)
Mood alteration-euphoria (Psychiatric disorders) | 1 (1)
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (muscle ache) (Musculoskeletal and connective tissue disorders) | 14 (21)
Nail changes (Skin and subcutaneous tissue disorders) | 37 (47)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 48 (132)
Nervous system disorders-Other, specify (vasovagal) (Nervous system disorders) | 1 (1)
Neurologic-Other (dizziness) (Nervous system disorders) | 3 (3)
Neuropathic pain (Nervous system disorders) | 6 (9) — e.g. jaw pain, neurologic pain, phantom pain , post-infectious neuralgia, or painful neuropathies
Neuropathy-sensory (Nervous system disorders) | 50 (88)
Neutrophil count decreased (Investigations) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 46 (142)
Ocular-Other (blurred vision) (Eye disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Pain-Other (dysethesia) (General disorders) | 17 (23)
Palpitation (Cardiac disorders) | 1 (1)
Partial thromboplastin time (PTT) (Investigations) | 10 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 1 (1)
Phlebitis (superficial) (Vascular disorders) | 4 (4)
Platelet count decreased (Investigations) | 3 (6)
Platelets (Investigations) | 27 (72)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Pericardial effusion/pericarditis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 11 (11)
Prothrombin time (PT) (Vascular disorders) | 5 (5)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 12 (13)
Renal/GU-Other (urgency) (Renal and urinary disorders) | 1 (1)
Rigors, chills (General disorders) | 9 (10)
Salivary gland changes (Gastrointestinal disorders) | 1 (1)
Sense of smell (Nervous system disorders) | 1 (1)
SGOT (AST) (Investigations) | 29 (48)
SGPT (ALT) (Investigations) | 19 (31)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin-Other (dry skin) (Skin and subcutaneous tissue disorders) | 2 (2)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Infections and infestations) | 10 (10)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT (Infections and infestations) | 9 (10)
Sweating (Skin and subcutaneous tissue disorders) | 5 (6)
Syncope (Nervous system disorders) | 2 (2)
Taste disturbance (dysgeusia) (Nervous system disorders) | 40 (86)
Tearing (watery eyes) (Eye disorders) | 3 (4)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrombosis/embolism (Vascular disorders) | 1 (1)
Transfusion:pRBCs (Blood and lymphatic system disorders) | 2 (3)
Tremor (Nervous system disorders) | 2 (3)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (6)
Tumor pain (onset or exacerbation of tumor pain due to treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ureteral obstruction (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 2 (3)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vision-blurred vision (Eye disorders) | 1 (1)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Voice changes/stridor/larynx (Respiratory, thoracic and mediastinal disorders) | 1 (2) — e.g. hoarseness, loss of voice, laryngitis
Vomiting (Gastrointestinal disorders) | 37 (66)
Weight loss (Investigations) | 17 (20)
White blood cell decreased (Investigations) | 5 (15)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Wound-infectious (Injury, poisoning and procedural complications) | 1 (1)
Wound-non-infectious (Injury, poisoning and procedural complications) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 19 (22)
Hypertension (Vascular disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No